

FreeSTyle LibRe and hospitAl admissions, morTality and qUality of life in high risk type 2 diabeteS patients (STRATUS study). Participant consent form.

Many thanks for taking the time to read about this study and for considering taking part. If you wish to be enrolled in the study please read the below statements carefully and initial in the boxes provided to show you are happy to continue.

| <ul> <li>I confirm that I have read the participant information sheet (version 1.6, 13.7.21) for the above study. I have had the opportunity to consider the information, ask questions and have had these answered satisfactorily.</li> <li>I understand that my participation is voluntary and that I am free to withdraw at any time without giving any reason, without my medical care or legal rights being affected.</li> <li>I understand that relevant sections of my medical notes and data collected during the study may be looked at by individuals from the study team, from the study sponsor (the University of Leeds) or by the NHS Trust. I give permission for these individuals to have access to my records.</li> <li>I understand that relevant sections of data collected during the study, may be looked at by individuals from the University, from</li> </ul> | | |
|---|---|---|
| regulatory authorities or from the NHS Trust, where it is relevant to my taking part in this research. I give permission for these individuals to have access to the research records. I understand that the information collected about me will be used to support other research in the future and may be shared anonymously with other researchers. No personal identifiable data will be shared. I agree for the study team to access my electronic patient records for the purpose of this study. I agree to my General Practitioner being informed of my participation in the study. I agree to take part in the above study. | | |
| Study site: | Participant study ID: | Date: |
| Participant full name: | Name of person taking consent: | Signature of consent taker: |
| Signature of participant: | | |
| Copy of consent form given to participant: YES/NO | | |